CLINICAL TRIAL: NCT02696057
Title: Bel-boyun ağrısı Nedeniyle başvuran Hastalarda farklı Fizyoterapi ve Manuel Terapi yöntemlerinin ağrı, Fonksiyon ve yaşam Kalitesi düzeyleri üzerin Etkisi
Brief Title: The Effect of Manual Therapy and Exercise in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GO13/550
Record Dates: First submitted 2016-02-24; First posted 2016-03-02 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual technics (Active Comparator): Manual technics was consisted of soft tissue technics, muscle energy technics, joint mobilization.
  Interventions: Other: manual technics
- Exercise (Active Comparator): Spinal stabilization exercises were applied all the patients in this group accompanied by physiotherapist.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: manual technics — soft tissue technics, joint mobilization and muscle energy technics were applied three sessions per week, totally six week.
  Arms: Manual technics
Other: Exercise — spinal stabilization exercise applied three sessions per week, totally six week.
  Arms: Exercise

SUMMARY:
Identification of the effects of spinal stabilization exercises and manual therapy methods on pain, function and quality of life in individuals with low back pain.

DETAILED DESCRIPTION:
113 patients participating in the study were divided into two groups. The patients in the physiotherapy group were instructed to perform special spinal stabilization exercises, while the patients in the manual therapy group were instructed to perform soft tissue mobilizations, muscle-energy techniques, joint mobilizations and/or manipulation methods depending on the nature of their lower back pain problems. Both groups were offered stabilization, strengthening, stretching, balance and exercise trainings as well as recommendations as to the daily life activities in line with the requirements of each individual. The severity of the pain suffered by the individuals was evaluated through a Visual Analog Scale. Oswestry Disability Index and Short Form-36 (SF-36) Scale were made respectively with respect to the functional condition and life quality. Assessments were repeated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic low back pain
* must have pain at least 3 or more according to Visual analog scale

Exclusion Criteria:

* Clinical diagnosis of Rheumatoid Arthritis
* Clinical diagnosis of Alzheimer
* Clinical diagnosis of Peripheral Neuropathy
* Clinical diagnosis of Diabetes Mellitus

Ages: 23 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
changes in pain severity | change from baseline in pain severity at 6 weeks.
  Visual Analog Scale:It is used in assessing the severity of pain. The scale is 10 cm long, which is labeled differently on each end (0= no pain, 10= the most severe pain)

SECONDARY OUTCOMES:
Changes of functional status | change from baseline in back functions at 6 weeks.
  Oswestry Disability Index: Various daily living activities are assessed by 10 questions each having a score of 0 to 5; points scored between 0 to 4 are recorded as no disability. Total score summed.
Changes in Quality of life | change form baseline in life quality levels at 6 weeks.
  SF-36 Quality of Life: this scale consists 36 item which assess pain, functional-emotional status, sleep, general health, mental health, social status and energy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PhD, Study Director — Hacettepe University; Ozlem Ulger, Asc. Proff, Principal Investigator — Hacettepe University; Seval Tamer, Msc, Study Director — Hacettepe University; Muzeyyen Oz, PT, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Health Sciences Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Slater SL, Ford JJ, Richards MC, Taylor NF, Surkitt LD, Hahne AJ. The effectiveness of sub-group specific manual therapy for low back pain: a systematic review. Man Ther. 2012 Jun;17(3):201-12. doi: 10.1016/j.math.2012.01.006. Epub 2012 Mar 3. PMID 22386046
- [Result] Steiger F, Wirth B, de Bruin ED, Mannion AF. Is a positive clinical outcome after exercise therapy for chronic non-specific low back pain contingent upon a corresponding improvement in the targeted aspect(s) of performance? A systematic review. Eur Spine J. 2012 Apr;21(4):575-98. doi: 10.1007/s00586-011-2045-6. Epub 2011 Nov 10. PMID 22072093
- [Result] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Result] Koes BW, Assendelft WJ, van der Heijden GJ, Bouter LM. Spinal manipulation for low back pain. An updated systematic review of randomized clinical trials. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2860-71; discussion 2872-3. doi: 10.1097/00007632-199612150-00013. PMID 9112710
- [Result] Dougherty PE, Karuza J, Savino D, Katz P. Evaluation of a modified clinical prediction rule for use with spinal manipulative therapy in patients with chronic low back pain: a randomized clinical trial. Chiropr Man Therap. 2014 Nov 18;22(1):41. doi: 10.1186/s12998-014-0041-8. eCollection 2014. PMID 25426289
- [Result] Huang SL, Liu YX, Yuan GL, Zhang J, Yan HW. Characteristics of lumbar disc herniation with exacerbation of presentation due to spinal manipulative therapy. Medicine (Baltimore). 2015 Mar;94(12):e661. doi: 10.1097/MD.0000000000000661. PMID 25816037
- [Result] Kosinski MR, Schein JR, Vallow SM, Ascher S, Harte C, Shikiar R, Frank L, Margolis MK, Vorsanger G. An observational study of health-related quality of life and pain outcomes in chronic low back pain patients treated with fentanyl transdermal system. Curr Med Res Opin. 2005 Jun;21(6):849-62. doi: 10.1185/030079905X46377. PMID 15969885